CLINICAL TRIAL: NCT02966236
Title: Impact of Tranexamic Acid Use in Transfusion Rate in Patients With Complex Kidney Stone Undergoing Percutaneous Nephrolithotomy: Randomised, Double-blind, Placebo Controlled Trial
Brief Title: Impact of Tranexamic Acid Use in Percutaneous Nephrolithotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Carlos Alfredo Batagello, PhD student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TXA
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Nephrolithiasis; Staghorn Calculus
Keywords: percutaneous nephrolithotomy
MeSH Terms: conditions — Nephrolithiasis; Staghorn Calculi | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid Group (Experimental): Tranexamic acid 1g IV during anesthesiology induction, single dose
  Interventions: Drug: Tranexamic Acid
- Placebo group (Placebo Comparator): normal saline 1g IV during anesthesiology induction, single dose
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic Acid Group
Drug: Placebos
  Arms: Placebo group

SUMMARY:
This study is a double blinded randomized controlled trial evaluating the impact of tranexamic acid use on the transfusion rate in patients with complex kidney stones undergoing percutaneous nephrolithotomy.

DETAILED DESCRIPTION:
Introduction: Kidney stone is a high incidence and prevalent disease affecting people around the world. Nearly 1 in 11 individuals in the United States will be affected at some point in their lives. Furthermore, stones are likely to recur with at least 50% of individuals experiencing another stone within 10 years of the first occurrence. Moreover, the disease mainly affects the economically active segment of the population with special social and economic implications in health.

Approximately 85% of stones are composed predominantly by calcium compounds and about 7% are attributed to urinary tract infections, named struvite stones, that usually develop as jagged structures called "staghorns" and can grow to be quite large, therefore becoming complex kidney stone. However, in HCFMUSP, as a Brazilian national reference center in urolithiasis treatment, this complex stones represents about 30 percent of all renal lithiasis treated.

This complex stones require individualized and specialized treatment, with percutaneous nephrolithotomy (PCNL) as the standard of care, with advantages of higher stone clearance and cost-effectiveness when compared with other treatment alternatives.

However, PCNL is associated with significant morbidity such as fever, urinary infections, septicemia and bleeding that may require blood transfusion. Of these complications bleeding is the most unpredictable and dreaded, and can lead to significant morbidity, beyond the potential risks of blood transfusions by itself.

In this way antifibrinolytic drugs, such as tranexamic acid, have been shown to reduce blood loss in a variety of surgical procedures, blood transfusion rate, morbidity and mortality related to bleeding.

Objectives: The main outcome measure of our study is to evaluate the impact of tranexamic acid use in blood transfusion rate in patients with complex kidney stones undergoing PCNL (number of patients receiving blood transfusions from surgery until hospital discharge). The secondary outcome is to evaluate blood loss by hemoglobin measure, surgical time, stone free rate and complications. Furthermore, we want to corroborate the drug safety, previously established in the medical literature.

Methods: After protocol approval by the hospital ethics committee, patients undergoing PCNL for complex renal stone (GUYS classification III and IV) and who provided written informed consent, will be eligible for the trial. After the patients' eligibility is confirmed, we will randomly allocate them to the intervention or placebo group by a computer program. Trial participants, care providers, surgeons, the anesthesiology team and data collectors will be blinded to group assignments. Patients will be managed with surgical standardized technique by Endourological HCFMUSP group and controlled care after surgery. Blood transfusion rate, hemoglobin drop and complications will be evaluated at 7, 30, 90 and 180 days after surgery. On postoperative day one, CT scan will be performed to assess stone free rate and complications.

ELIGIBILITY:
Inclusion Criteria:

* Complex kidney stone (staghorn calculi GUYS III and IV)

Exclusion Criteria:

* Coronary artery disease - stent
* Severe chronic renal failure
* Congenital or acquired thrombophilia/thrombosis event
* Known or suspected allergy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
blood transfusion rate | two years
  postoperative follow up

SECONDARY OUTCOMES:
blood loss | two years
  postoperative follow up
surgical time | two years
  postoperative follow up
stone free rate | two years
  postoperative follow up
complications | two years
  postoperative follow up

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo Medical School, São Paulo, Brazil

REFERENCES:
- [Derived] Batagello CA, Vicentini FC, Monga M, Miller AW, Marchini GS, Torricelli FCM, Danilovic A, Coelho RF, Srougi M, Nahas WC, Mazzucchi E. Tranexamic acid in patients with complex stones undergoing percutaneous nephrolithotomy: a randomised, double-blinded, placebo-controlled trial. BJU Int. 2022 Jan;129(1):35-47. doi: 10.1111/bju.15378. Epub 2021 Jun 13. PMID 33630393